CLINICAL TRIAL: NCT05808530
Title: The Effect of Cognitive Stimulation Therapy on Apathy, Loneliness, Anxiety and Activities of Daily Living in Elderly Individuals Diagnosed With Alzheimer's
Brief Title: Cognitive Stimulation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Eda Atay, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Hasan Kalyoncuuuu University
Record Dates: First submitted 2023-01-14; First posted 2023-04-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease 10; Dementia; Apathy; Anxiety; Loneliness
Keywords: Alzheimer Disease; Dementia; Apathy; Anxiety; Loneliness; Cognitive Stimulation Therapy
MeSH Terms: conditions — Alzheimer Disease 10; Dementia; Lethargy; Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): It is te intervention grup.
  Interventions: Behavioral: Cognitive Stimulation Therapy
- no intervention arm (No Intervention): It is the non intervention group.

INTERVENTIONS:
Behavioral: Cognitive Stimulation Therapy — CST involves the use of standard tasks that focus on cognitive functions, designed to meet varying levels of difficulty in accordance with the individual's ability and rehabilitation. A detailed guide for CST is available for a range of health and care professionals, including care workers, occupational therapists, psychologists, and nurses (https://www.ucl.ac.uk/international-cognitive-stimulation-therapy/) publications/cst-manuals). The CST application consists of 14 sessions of 45-50 minutes, 2 days a week.
  Intervention Group Week 1=Getting acquainted and applying pre-tests Week 2=Physical games and Sounds Week 3=Childhood and Food Week 4=Current events and Faces / Scenes Week 5=Word association and Creativity Week 6=Categorizing Objects and Orientation Week 7= Money usage and Games Week 8=Word Games and Team Competition Week 9=Closing and post-test application
  Arms: Intervention arm

SUMMARY:
The concept of cognitive stimulation in AD is one of the most popular approaches. Cognitive Stimulation Therapy (CST) is stated to be evidence-based best practice with robust clinical trials, administered according to specific guidelines for individuals with mild to moderate dementia. In this study, it was aimed to investigate the effects of CST application on the levels of apathy, loneliness, anxiety and daily living activities in elderly individuals with Alzheimer's disease.

This research was planned in an experimental research design with a single center and pretest posttest control group. The research was planned to be carried out between January 2023 and June 202 at the Moral House of Gaziantep Metropolitan Municipality, Department of Disabled and Health Services. Introductory Information Form, Standardized Mini-Mental Test, Geriatric Anxiety Scale, Apathy Rating Scale, Loneliness Scale and Functional Disability in Dementia Scale will be used in the research. CST will be administered by a researcher trained in therapy, 2 days a week, for a total of 14 sessions of 45-50 minutes. There will be a pre-test before the application, an intermediate test right after the application, and a post-test three months later. Research data will be evaluated in SPSS 25.0 New York package program.

DETAILED DESCRIPTION:
Alzheimer's Disease is an insidious onset and slowly progressive disease, characterized by the presence of cognitive, behavioral and general dysfunction. Among the neuropsychiatric and behavioral symptoms seen in Alzheimer's patients, apathy is the most common symptom. It is also followed by depression, aggression, anxiety and sleep disorders. Behavioral and psychological symptoms (BPSD) affect up to 90% of people with dementia during the illness. Therefore, it brings great difficulties to both patients and their caregivers and causes low quality of life. In addition, the inability to treat the disease completely worsens this situation. Considering the pharmacological treatment of psychological symptoms such as apathy, anxiety, depression in AD individuals, the existence of adverse side effects, increased mortality, limited drug efficacy, relatively high cost, and the inability to effectively treat some of the most distressing behaviors, it is recommended to give priority to non-pharmacological interventions.

The concept of cognitive stimulation in AD is one of the most popular approaches. It is stated that Cognitive Stimulation Therapy (CST) is the best evidence-based practice with robust clinical trials, applied according to a specific guideline for individuals with mild and moderate dementia. In addition, CST is the only intervention recommended by the UK's National Institute for Clinical Excellence (NICE) to promote cognition, independence and well-being for people with mild to moderate dementia. It has been determined that CST has many effects on individuals with Alzheimer's disease. However, there are different results in studies on the effectiveness of cognitive intervention strategies aimed at reducing cognitive functions, behavioral and psychiatric symptoms. To enable the conversion of CST into routine clinical practice, practice research to support the standardization and generalization of cognitive stimulation therapy planned for patients with AD and its impact on improving neuropsychiatric symptoms and daily living skills requires further research. In addition, the absence of a widely used standard guideline for pharmacological methods for patients with AD in our country reveals that the planned study will contribute to practice. It has been confirmed by many studies that CST applied to individuals with AD contributes to the strengthening of cognitive, psychological and social aspects, but there are few studies applied by nurses. It is noteworthy that the studies on the CST program applied by nurses in our country are limited. Therefore, the need for more clinical studies is emphasized by nurses to build and disseminate knowledge in this area, as the intervention has been little studied. In addition, the absence of a widely used standard guideline for pharmacological methods for patients with AD in our country reveals that the planned study will contribute to practice. In this study, it is aimed to investigate the effect of CST application on the levels of apathy, loneliness, anxiety and daily living activities in elderly individuals diagnosed with Alzheimer's.

This research was planned in a single center and experimental research design with pretest posttest control group. The research was planned to be carried out between January 2023 and June 202 at the Moral House affiliated to Gaziantep Metropolitan Municipality Disabled and Health Services Department. Introductory Information Form, Standardized Mini-Mental Test, Geriatric Anxiety Scale, Apathy Rating Scale, Loneliness Scale and Functional Disability in Dementia Scale will be used in the research. CST will be applied by a trained researcher in therapy, 2 days a week, in a total of 14 sessions of 45-50 minutes. There will be a pre-test before the application, an intermediate test right after the application, and a post-test three months later. Research data will be evaluated in SPSS 25.0 New York package program.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older,
* Having a mild Alzheimer's diagnosis and a Standardized Mini Mental Test score in the range of 18-23,
* Able to speak and understand Turkish,
* Hearing, understanding, seeing and speaking problems,
* Having no physical illness or disability to participate in group work,
* Have not participated in the CST program before, Individuals who volunteer to participate in the research will be included in the study.

Exclusion Criteria:

* Not meeting any of the research inclusion criteria,
* Have not attended at least two sessions of the CST program,
* Patients who refuse/want to leave the CST program will be excluded from the study by the investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The effect of CST on the level of apathy in Alzheimer's patients | through study completion, an average of 1 year
  The level of apathy will be measured withAphaty Evaluation Scale in Alzheimer's patients after CST.
The effect of CST on the level of loneliness in Alzheimer's patients | through study completion, an average of 1 year
  The level of loneliness will be measured with a UCLA Loneliness Scale in Alzheimer's patients after CST.
The effect of CST on the level of anxiety in Alzheimer's patients | through study completion, an average of 1 year
  The level of anxiety will be measured with a Geraitric Anxiety Scale in Alzheimer's patients after CST.
The effect of CST on the level of Activities of Daily Living in Alzheimer's patients | through study completion, an average of 1 year
  The level of anxiety will be measured with a Activities of Daily Living Scale in Alzheimer's patients after CST.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juarez-Cedillo T, Gutierrez-Gutierrez L, Sanchez-Hurtado LA, Martinez-Rodriguez N, Juarez-Cedillo E. Randomized Controlled Trial of Multi-Component Cognitive Stimulation Therapy (SADEM) in Community-Dwelling Demented Adults. J Alzheimers Dis. 2020;78(3):1033-1045. doi: 10.3233/JAD-200574. PMID 33104028
- [Background] Zhao QF, Tan L, Wang HF, Jiang T, Tan MS, Tan L, Xu W, Li JQ, Wang J, Lai TJ, Yu JT. The prevalence of neuropsychiatric symptoms in Alzheimer's disease: Systematic review and meta-analysis. J Affect Disord. 2016 Jan 15;190:264-271. doi: 10.1016/j.jad.2015.09.069. Epub 2015 Oct 24. PMID 26540080
- [Background] Cerejeira J, Lagarto L, Mukaetova-Ladinska EB. Behavioral and psychological symptoms of dementia. Front Neurol. 2012 May 7;3:73. doi: 10.3389/fneur.2012.00073. eCollection 2012. PMID 22586419
- [Background] Sobral SR, Sobral M. Computerized cognitive stimulation for people with dementia or with mild cognitive impairment: a bibliometric review. Dement Neuropsychol. 2021 Jan-Mar;15(1):28-40. doi: 10.1590/1980-57642021dn15-020003. PMID 33907595
- [Background] Perkins L, Fisher E, Felstead C, Rooney C, Wong GHY, Dai R, Vaitheswaran S, Natarajan N, Mograbi DC, Ferri CP, Stott J, Spector A. Delivering Cognitive Stimulation Therapy (CST) Virtually: Developing and Field-Testing a New Framework. Clin Interv Aging. 2022 Feb 9;17:97-116. doi: 10.2147/CIA.S348906. eCollection 2022. PMID 35173425
- [Background] Fukushima RLM, do Carmo EG, Pedroso RDV, Micali PN, Donadelli PS, Fuzaro G Junior, Venancio RCP, Viola J, Costa JLR. Effects of cognitive stimulation on neuropsychiatric symptoms in elderly with Alzheimer's disease: A systematic review. Dement Neuropsychol. 2016 Jul-Sep;10(3):178-184. doi: 10.1590/S1980-5764-2016DN1003003. PMID 29213453
- [Background] Khan Z, Corbett A, Ballard C. Cognitive stimulation therapy: training, maintenance and implementation in clinical trials. Pragmat Obs Res. 2014 Apr 5;5:15-19. doi: 10.2147/POR.S56000. eCollection 2014. PMID 27774025
- [Background] Wong GHY, Yek OPL, Zhang AY, Lum TYS, Spector A. Cultural adaptation of cognitive stimulation therapy (CST) for Chinese people with dementia: multicentre pilot study. Int J Geriatr Psychiatry. 2018 Jun;33(6):841-848. doi: 10.1002/gps.4663. Epub 2017 Jan 11. PMID 29717527
- [Background] Yang YP, Lee FP, Chao HC, Hsu FY, Wang JJ. Comparing the Effects of Cognitive Stimulation, Reminiscence, and Aroma-Massage on Agitation and Depressive Mood in People With Dementia. J Am Med Dir Assoc. 2016 Aug 1;17(8):719-24. doi: 10.1016/j.jamda.2016.03.021. Epub 2016 May 7. PMID 27168052
- [Background] Hall L, Orrell M, Stott J, Spector A. Cognitive stimulation therapy (CST): neuropsychological mechanisms of change. Int Psychogeriatr. 2013 Mar;25(3):479-89. doi: 10.1017/S1041610212001822. Epub 2012 Nov 12. PMID 23146408
- [Background] Chen HM, Tsai LJ, Chao SY, Clark MJ. Study on the Effects of Individualized Learning Therapy on Cognitive Function and Behavioral and Psychological Symptoms of Dementia in the Institutionalized Older Adults. J Nurs Res. 2016 Dec;24(4):300-310. doi: 10.1097/JNR.0000000000000118. PMID 27846102
- [Background] Lin HC, Yang YP, Cheng WY, Wang JJ. Distinctive effects between cognitive stimulation and reminiscence therapy on cognitive function and quality of life for different types of behavioural problems in dementia. Scand J Caring Sci. 2018 Jun;32(2):594-602. doi: 10.1111/scs.12484. Epub 2017 Sep 7. PMID 28881430
- [Background] Lok N, Buldukoglu K, Barcin E. Effects of the cognitive stimulation therapy based on Roy's adaptation model on Alzheimer's patients' cognitive functions, coping-adaptation skills, and quality of life: A randomized controlled trial. Perspect Psychiatr Care. 2020 Jul;56(3):581-592. doi: 10.1111/ppc.12472. Epub 2020 Jan 12. PMID 31930518
- [Background] Martinez-Moreno M, Cerulla N, Chico G, Quintana M, Garolera M. Comparison of neuropsychological and functional outcomes in Alzheimer's disease patients with good or bad response to a cognitive stimulation treatment: a retrospective analysis. Int Psychogeriatr. 2016 Nov;28(11):1821-1833. doi: 10.1017/S104161021600123X. Epub 2016 Aug 9. PMID 27503001